CLINICAL TRIAL: NCT00833963
Title: An Observational Study of Pregnancy and Pregnancy Outcomes in Women With Breast Cancer Treated With Herceptin, Perjeta in Combination With Herceptin, or Kadcyla During Pregnancy or Within 7 Months Prior to Conception
Brief Title: A Study of Pregnancy and Pregnancy Outcomes in Women With Breast Cancer Treated With Trastuzumab, Pertuzumab in Combination With Trastuzumab, or Ado-Trastuzumab Emtansine
Acronym: MotHER
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: H4621g
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Pregnancy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants Treated With Trastuzumab: Participants who are being treated with trastuzumab during pregnancy or within 7 months prior to conception will be evaluated for cancer and pregnancy as determined by their treating physicians' standards of care, and will be observed for up to 12 months after delivery.
  Interventions: Drug: Trastuzumab
- Participants Treated With Trastuzumab and Pertuzumab: Participants who are being treated with the combination of trastuzumab and pertuzumab during pregnancy or within 7 months prior to conception will be evaluated for cancer and pregnancy as determined by their treating physicians' standards of care, and will be observed for up to 12 months after delivery.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Participants Treated With Ado-Trastuzumab Emtansine: Participants who are being treated with ado-trastuzumab emtansine during pregnancy or within 7 months prior to conception will be evaluated for cancer and pregnancy as determined by their treating physicians' standards of care, and will be observed for up to 12 months after delivery.
  Interventions: Drug: Ado-Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab — Participants will receive trastuzumab as determined by their treating physicians' standards of care.
  Other Names: Herceptin
  Groups: Participants Treated With Trastuzumab; Participants Treated With Trastuzumab and Pertuzumab
Drug: Pertuzumab — Participants will receive pertuzumab as determined by their treating physicians' standards of care.
  Other Names: Perjeta
  Groups: Participants Treated With Trastuzumab and Pertuzumab
Drug: Ado-Trastuzumab Emtansine — Participants will receive ado-trastuzumab emtansine as determined by their treating physicians' standards of care.
  Other Names: Kadcyla
  Groups: Participants Treated With Ado-Trastuzumab Emtansine

SUMMARY:
The MotHER Pregnancy Registry is a United States (U.S.)-based, prospective, observational cohort study in women with breast cancer who have been or are being treated with a trastuzumab (herceptin)-containing regimen with or without pertuzumab (perjeta) or ado-trastuzumab emtansine (kadcyla) during pregnancy or within 7 months prior to conception (regardless of cancer stage at the time of trastuzumab, pertuzumab, or ado-trastuzumab emtansine exposure).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant; women identified at any trimester of pregnancy may enroll in this study as long as enrollment occurs prior to experiencing pregnancy outcome (that is [i.e.], live birth, stillbirth, or abortion)
* Exposure to at least one dose of trastuzumab (as adjuvant or metastatic treatment), pertuzumab plus trastuzumab combination treatment, or ado-trastuzumab emtansine during pregnancy or within 7 months prior to conception
* United States resident

Exclusion Criteria:

* Prior knowledge of pregnancy outcome (i.e., live birth, stillbirth, or abortion) at time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is recruiting participants from anywhere within the United States. No office visits are required to participate in this registry. Information is collected from participants based on their medical charts.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01-14 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants Developing Oligohydramnios | From enrollment up to the delivery or upon termination of pregnancy (up to 12 months)
Number of Live Births | From Week 20 of gestation to the delivery or upon termination of pregnancy (up to 12 months)
Number of Fetal Deaths/Stillbirths | From Week 20 of gestation to the delivery or upon termination of pregnancy (up to 12 months)
Number of Fetal or Infant Major Malformations | From delivery up to 12 months after delivery
Number of Fetal or Infant Deformations | From delivery up to 12 months after delivery
Number of Fetal or Infant Disruptions | From delivery up to 12 months after delivery
Number of Fetal or Infant Functional Deficits | From delivery up to 12 months after delivery

SECONDARY OUTCOMES:
Number of Spontaneous Abortions | From enrollment up to 12 months
Number of Therapeutic Abortions, or Elective Abortions | From enrollment up to 12 months
Number of Premature Births | From enrollment up to 12 months
Number of Infants Small for Gestational Age | From delivery up to 12 months after delivery
Number of Cases of Intrauterine Growth Restriction (IUGR) | From enrollment up to 12 months
Number of Other Specific Pregnancy or Delivery Complications | From enrollment up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vikki Brown, M.D., Study Director — Syneos Health
Locations (1):
- Kendle International, Inc, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Perachino M, Poggio F, Arecco L, Blondeaux E, Spinaci S, Marrocco C, Levaggi A, Lambertini M. Update on Pregnancy Following Breast Cancer Diagnosis and Treatment. Cancer J. 2022 May-Jun 01;28(3):176-182. doi: 10.1097/PPO.0000000000000599. PMID 35594464